CLINICAL TRIAL: NCT05283590
Title: Automated Inferior Vena Cava Collapsibility Index for Assessing Fluid Responsiveness in Ventilated Patients After Cardiac Surgery.
Brief Title: Automated Inferior Vena Cava Collapsibility Index Fluid Responsiveness in Ventilated Patients After Cardiac Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-21-947
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-02

CONDITIONS: Hemodynamic Monitoring; ICU; Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: The IVC will be measured by the automated mode and manual measures will be recorded. All patients will have PPv by LiDCO
  Interventions: Diagnostic Test: Automated echocardiographic inferior vena cava measurement

INTERVENTIONS:
Diagnostic Test: Automated echocardiographic inferior vena cava measurement — Patients will be place in supine position. view: subcostal view, importantly supine is standard position for IVC measurement, the IVC is larger in the right lateral decubitus position and vice versa, alternatively directly through a transhepatic approach. Measures will be performed in the two dimensional mode close to the hepatic vein (1 - 3cm from the IVC connection to the right atrium). The IVC will be measured by MM-Mode manually and with the automated mode (both measures will be recorded. In the manual mode this measure requires concurrent utilization of M-Mode and two dimensional mode
  Other Names: Manual echocardiographic inferior vena cava measurement; LiDCO

SUMMARY:
Echocardiographic measurement of inferior vena cava (IVC) collapsibility index (CI) with automated software analyses has been introduced. This study aims to assess the accuracy of IVC-CI (caval index) measurements as well as the ability to track fluid responsiveness (FRes) over time comparing the automated echocardiographic method with the pulse pressure variation (PPV) technique and the manual echocardiographic method in cardiac surgery patients.

DETAILED DESCRIPTION:
It is expected to have insights about the concordance rate. The automated echocardiographic method of measuring CI method may or may not meet the criteria for interchangeability with the thermodilution technique or the manual echocardiographic method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age more than18 years old. 2. Cardiac surgical patients including (coronary artery bypass graft surgery, valvular surgeries, and aortic dissection surgeries) 3. Need for decision to administer IV fluids (hypotension that require assessment and possible fluid boluses defined as a systolic blood pressure less than 90mmHg. Normotensive patients who require fluid therapy with any other manifestation of low perfusion including tachycardia, low urine output, increased core-peripheral temperature gradient, serial increase in serum lactate, and serial increase in base deficit, and normotensive). The endpoint of fluid resuscitation is return normal blood pressure

Exclusion Criteria:

-1. Contraindication for fluid administration including acute pulmonary edema. 2. Moderate or more tricuspid valve lesion or pulmonary hypertension (more 50 mmHg) where high central venous pressure is expected 3. Patients on hemodialysis. 4. Patient on intra-aortic balloon pump (IABP) or extracorporeal membrane oxygenation (ECMO) 5. Irregular cardiac rhythm: patients with atrial fibrillation or frequent ectopics are excluded.

6. Patients with chest open 7. Poor echocardiography window (The images will be stored and analyzed by senior physician within the ICU certified in echocardiography)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective, descriptive, single-center study that will examine three techniques for guiding fluid therapy. Patients who are in need of fluid therapy will be identified. The study will be conducted over one year after the approval of the ethical committee. Patients after cardiac surgery will be recuited
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness rate 500cc of colloids over 10 min. | 30 minutes
  defined as increase in the stoke volume by 15% after infusion of 500cc of colloids

SECONDARY OUTCOMES:
HR | 30 minutes
  before and after the fluid challenge
MAP | 30 minutes
  before and after the fluid challenge
VTI | 30 minutes
  before and after the fluid challenge

CONTACTS AND LOCATIONS:
Overall Officials: Amr Omar, Md, PhD, Principal Investigator — Hamad medical corproation
Locations (1):
- Hamad medical corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
No allowed by our corporate